CLINICAL TRIAL: NCT05137054
Title: Phase 1b Study of REGN5458 (Anti-BCMA x Anti-CD3 Bispecific Antibody) Plus Other Cancer Treatments for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Examine the Effects of Novel Therapy Linvoseltamab in Combination With Other Cancer Treatments for Adult Patients With Multiple Myeloma That is Resistant to Current Standard of Care Treatments
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2012; 2020-004638-39 (EudraCT Number); 2023-506247-42-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-11-18; First posted 2021-11-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma (RRMM); B-cell maturation antigen (BCMA); Anti-CD3 monoclonal antibodies (mAbs)
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; carfilzomib; Lenalidomide; Bortezomib; pomalidomide; isatuximab; cemiplimab; nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Linvoseltamab + Daratumumab (Experimental): Linvoseltamab + Daratumumab
  Interventions: Drug: Linvoseltamab; Drug: Daratumumab
- Cohort 2: Linvolseltamab + Carfilzomib (Experimental): Linvoseltamab + Carfilzomib
  Interventions: Drug: Linvoseltamab; Drug: Carfilzomib
- Cohort 3: Linvoseltamab + Lenalidomide (Experimental): Linvoseltamab + Lenalidomide
  Interventions: Drug: Linvoseltamab; Drug: Lenalidomide
- Cohort 4: Linvoseltamab + Bortezomib (Experimental): Linvoseltamab + Bortezomib
  Interventions: Drug: Linvoseltamab; Drug: Bortezomib
- Cohort 5: Linvoseltamab + Pomalidomide (Experimental): Linvoseltamab + Pomalidomide
  Interventions: Drug: Linvoseltamab; Drug: Pomalidomide
- Cohort 6: Linvoseltamab + Isatuximab (Experimental): Linvoseltamab + Isatuximab
  Interventions: Drug: Linvoseltamab; Drug: Isatuximab
- Cohort 7: Linvoseltamab + Fianlimab (Experimental): Linvoseltamab + Fianlimab
  Interventions: Drug: Linvoseltamab; Drug: Fianlimab
- Cohort 8: Linvoseltamab + Cemiplimab (Experimental): Linvoseltamab + Cemiplimab
  Interventions: Drug: Linvoseltamab; Drug: Cemiplimab
- Cohort 9: Linvoseltamab + Nirogacestat (Experimental): Linvoseltamab + Nirogacestat
  Interventions: Drug: Linvoseltamab; Drug: Nirogacestat
- Cohort 10: Linvoseltamab + Cevostamab (Experimental): Linvoseltamab + Cevostamab
  Interventions: Drug: Linvoseltamab; Drug: Cevostamab

INTERVENTIONS:
Drug: Linvoseltamab — Linvoseltamab is administered by intravenous (IV) infusion
  Other Names: REGN5458; Lynozyfic™
Drug: Daratumumab — Daratumumab is administered by IV infusion and/or subcutaneous (SC) injection; SC injection may be used after a minimum of 2 cycles of IV administration at the investigator's discretion.
  Other Names: Darzalex®; Darzalex Faspro™
  Arms: Cohort 1: Linvoseltamab + Daratumumab
Drug: Carfilzomib — Carfilzomib is administered by IV infusion
  Other Names: Kyprolis®
  Arms: Cohort 2: Linvolseltamab + Carfilzomib
Drug: Lenalidomide — Lenalidomide is administered by mouth (PO) as a capsule
  Other Names: Revlimid®
  Arms: Cohort 3: Linvoseltamab + Lenalidomide
Drug: Bortezomib — Bortezomib is administered by IV infusion or SC injection
  Other Names: Velcade®
  Arms: Cohort 4: Linvoseltamab + Bortezomib
Drug: Pomalidomide — Pomalidomide is administered by mouth (PO) as a capsule
  Other Names: Imnovid, Pomalyst®
  Arms: Cohort 5: Linvoseltamab + Pomalidomide
Drug: Isatuximab — Isatuximab is administered by IV infusion
  Other Names: Sarclisa®
  Arms: Cohort 6: Linvoseltamab + Isatuximab
Drug: Fianlimab — Fianlimab is administered by IV infusion
  Other Names: REGN3767
  Arms: Cohort 7: Linvoseltamab + Fianlimab
Drug: Cemiplimab — Cemiplimab is administered by IV infusion
  Other Names: LIBTAYO; REGN2810
  Arms: Cohort 8: Linvoseltamab + Cemiplimab
Drug: Nirogacestat — Nirogacestat is administered by mouth (PO) as a tablet
  Other Names: PF-03084014
  Arms: Cohort 9: Linvoseltamab + Nirogacestat
Drug: Cevostamab — Cevostamab is administered by IV infusion
  Other Names: BFCR4350A; RO7187797
  Arms: Cohort 10: Linvoseltamab + Cevostamab

SUMMARY:
This study is researching an experimental drug called linvoseltamab in combination with other drugs for the treatment of a blood cancer called multiple myeloma. Linvoseltamab has previously been studied as a single agent (without other cancer treatments) in participants with multiple myeloma that returned after prior therapies and needed to be treated again.

In the initial study, some participants treated with linvoseltamab had improvement of their myeloma, including complete responses (no evidence of myeloma in their bodies).

This study is the first time linvoseltamab will be combined with other cancer therapies.

The main goal is to understand if linvoseltamab can be given safely with other cancer treatments, and if so, what dose of linvoseltamab should be used for each combination.

The study is looking at several other research questions, including:

* How many participants treated with linvoseltamab in combination with each of the other cancer treatments have improvement of their multiple myeloma
* What side effects may happen from taking linvoseltamab together with another cancer treatment
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug(s) (which could make the study drug(s) less effective or could lead to side effects)

ELIGIBILITY:
General Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
2. Participants must have measurable disease as defined in the protocol according to International Myeloma Working Group (IMWG) consensus criteria
3. Adequate creatinine clearance, hematologic function and hepatic function, as defined in protocol
4. Life expectancy of at least 6 months.

Cohort Specific Inclusion Criteria:

For cohorts 1-6, each participant must have RRMM with progression following at least 3 lines of therapy, or at least 2 lines of therapy and either prior exposure to at least 1 anti-CD38 antibody, 1 immunomodulatory imide drug (IMiD) and 1 proteasome inhibitor (PI), or double-refractory to 1 PI and 1 IMiD, or the combination of 1 PI and 1 IMiD.

Cohort 1: Prior treatment with daratumumab is allowed if previously tolerated. However, participants enrolled in the expansion portion cannot be refractory to an anti-CD38 antibody containing regimen. In addition, all participants must have at least a 6-month washout from prior anti-CD38 antibody therapy.

Cohort 2: Prior treatment with carfilzomib is allowed if previously tolerated at the approved full dose. Carfilzomib-refractory participants may enroll in the dose finding portion provided they are triple-class refractory (PI, IMiD, anti-CD38 antibody). However, participants enrolled in the dose expansion portion cannot be refractory to carfilzomib. In addition, all participants must have at least a 6-month washout from prior carfilzomib therapy.

Cohort 3: Prior treatment with lenalidomide is allowed if previously tolerated at the approved full dose. However, a participant cannot be refractory to any combination regimen that included 25 mg of lenalidomide. In addition, participants must have at least a 6-month washout from any prior lenalidomide therapy (including maintenance therapy).

Cohort 4: Prior treatment with bortezomib is allowed if previously tolerated at the approved full dose. Bortezomib-refractory participants may enroll in the dose finding portion provided they are triple-class refractory (PI, IMiD, anti-CD38 antibody). However, participants enrolled in the dose expansion portion cannot be refractory to bortezomib. In addition, all participants must have at least a 6-month washout from prior bortezomib therapy.

Cohort 5: Prior treatment with pomalidomide is allowed if previously tolerated at the approved full dose. Additionally, participants must undergo at least a 6-month washout following prior pomalidomide therapy before enrollment.

Cohort 6: Prior treatment with isatuximab is allowed if previously tolerated. Additionally, participants must undergo at least a 3-month washout following prior anti-CD38 antibody therapy before enrollment.

Cohort 7 and 8: RRMM with progressive disease and received at least 3 lines of therapy including exposure to at least 1 anti-CD38 antibody, 1IMiD, and 1 PI or triple-class refractory disease (anti-CD38 antibody, IMiD, PI).

Cohort 9: Progressive RRMM in participants with triple-class refractory disease (anti-CD38 antibody, IMiD, PI) after at least 3 lines of therapy Cohort 10: Progressive RRMM after at least 3 lines of therapy including exposure to at least 1 anti-CD38 antibody, 1 IMiD, and 1 PI.

General Key Exclusion Criteria:

1. Diagnosis of plasma cell leukemia, primary light-chain amyloidosis (excluding myeloma associated amyloidosis), Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
2. Participants with known MM brain lesions or meningeal involvement
3. Treatment with any systemic anti-myeloma therapy within 5 half-lives or within 21 days prior to first administration of study drug regimen, whichever is shorter
4. History of allogeneic and autologous stem cell transplantation, as described in the protocol
5. Unless stated otherwise in a specific sub-protocol, prior treatment with a T cell-based immunotherapy directed against BCMA bispecific antibodies and bispecific T-cell engagers (BiTEs), and BCMA chimeric antigen receptor (CAR) T cells (Note: BCMA antibody-drug conjugates are not excluded)
6. History of progressive multifocal leukoencephalopathy, neurodegenerative condition or central nervous system (CNS) movement disorder or participants with a history of seizure within 12 months prior to study enrollment are excluded
7. Live or attenuated vaccination within 28 days prior to first study drug regimen administration with a vector that has replicative potential
8. Cardiac ejection fraction <40% by echocardiogram (Echo) or multigated acquisition (MUGA) scan.

Cohort Specific Exclusion Criteria:

Cohort 2:

1. Dose expansion: Prior treatment with a B-cell maturation antigen (BCMA) -directed CAR T-cell therapy will not be exclusionary if completed at least 12 weeks prior to first study treatment

Cohort 3:

1. Known malabsorption syndrome or pre-existing gastrointestinal (GI) condition that may impair absorption of lenalidomide; delivery of lenalidomide via nasogastric tube or gastrostomy tube is not allowed.

Cohort 4:

1. Peripheral neuropathy grade ≥2

Cohort 5:

1. Known malabsorption syndrome or pre-existing GI conditions that may impair absorption of pomalidomide; delivery of pomalidomide via nasogastric tube or gastrostomy tube is not allowed.

Cohort 7:

1. Prior treatment with anti-lymphocyte activation gene 3 (LAG-3) agents. Prior exposure to vaccine therapies or other immune checkpoint modulating therapies such as anti-programmed cell death protein 1 (PD-1) antibodies is permitted, as described in the protocol.
2. Ongoing or recent (within 2 years) evidence of an autoimmune disease that has required systemic treatment with immunosuppressive agents, as described in the protocol.
3. Prior solid organ transplant.
4. History of grade ≥3 immune-mediated adverse events (with the exclusion of endocrinopathies that are fully controlled by hormone replacement) from prior checkpoint inhibitor therapies.

Cohort 8:

1. Prior treatment with anti-PD-1 or anti-PD-L1 agents. Prior exposure to vaccine therapies or other immune checkpoint modulating therapies such as anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibodies is permitted, as described in the protocol.
2. Encephalitis or meningitis in the year prior to enrollment.
3. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years. A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥6 months prior to enrollment.
4. Ongoing or recent (within 2 years) evidence of an autoimmune disease that has required systemic treatment with immunosuppressive agents, as described in the protocol.
5. Prior solid organ transplant.
6. History of grade ≥3 immune-mediated adverse events (with the exclusion of endocrinopathies that are fully controlled by hormone replacement) from prior checkpoint inhibitor therapies.

Cohort 9:

1. Abnormal QT interval corrected by Fridericia's formula (QTcF), as described in the protocol
2. Use of concomitant medications that are known to prolong the QT/QTcF interval including Class Ia and Class III antiarrhythmics at the time of informed consent
3. Ongoing use or anticipated use of food or drugs that are known strong/moderate cytochrome P450 (CYP)3A4 inhibitors, or strong CYP3A inducers within 14 days prior to first dose of nirogacestat
4. Known malabsorption syndrome or existing gastrointestinal GI condition that may impair absorption of nirogacestat; delivery of nirogacestat via nasogastric tube or gastrostomy tube is not allowed.

Cohort 10:

1. Known or suspected active Epstein-Barr virus (EBV) infection.
2. Known history of Hemophagocytic lymphohistiocytosis/Macrophage activation syndrome (HLH/MAS).
3. Prior treatment with cevostamab or another agent with the same target [Fragment crystallizable receptor-like 5 (FcRH5)].

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2028-04-11 (Estimated); Study Completion 2034-09-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of pre-defined safety criteria or dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period | Up to 28 Days
  Dose finding portion only
Incidence of treatment-emergent adverse events (TEAEs) | Up to 5 Years
Severity of TEAEs | Up to 5 Years
Incidence of serious adverse events (SAEs) | Up to 5 Years
Severity of SAEs | Up to 5 Years
Incidence of adverse events of special interest (AESIs) | Up to 5 Years
Severity of AESIs | Up to 5 Years
Incidence of laboratory abnormalities | Up to 5 Years
  ≥ grade 3 per National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE v5.0]

SECONDARY OUTCOMES:
Objective response rate (ORR) as measured by International Myeloma Working Group (IMWG) criteria | Up to 5 Years
Duration of response (DOR) by IMWG criteria | Up to 5 Years
Progression-free survival (PFS) as measured by IMWG criteria | Up to 5 Years
Rate of minimal residual disease (MRD) negative status by IMWG criteria | Up to 5 Years
Concentrations of total linvoseltamab in serum over time | Up to 5 Years
Incidence over time of anti-drug antibodies (ADAs) to linvoseltamab | Up to 5 Years
Overall Survival (OS) | Up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (42):
- United States (13):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Health Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medicine/New York Presbyterian Hospital, New York, New York
  - New York Presbyterian Hospital Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - VA Puget Sound Health Care System, Seattle, Washington
- France (10):
  - CHU de Lille - Rue Michel Polonovski, Lille, Nord
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers, Nouvelle-Aquitaine
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire Angers, Angers
  - CHU Montpellier - Departement D'Hematologie, Montpellier
  - Saint Antoine Hospital, Paris
  - Institut Gustave Roussy, Villejuif
  - Hospital Henri Mondor, Créteil, Île-de-France Region
  - Saint Louis Hospital, Paris, Île-de-France Region
  - Hopital Necker, Paris, Île-de-France Region
- Greece (2):
  - Evangelismos General Hospital, Athens, Attica
  - General Hospital of Athens Alexandra, Athens
- Israel (3):
  - Sheba Medical Center, Ramat Gan, Central District
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
- Spain (14):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia (ICO) - Hospital Duran i Reynals,, Barcelona
  - Universitaru Hospital La Princesa, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Psiquiatria, Madrid
  - University Hospital and Research Institute, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - University Hospital of Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/